CLINICAL TRIAL: NCT06115226
Title: Laparascopic vs. Laparotomy Management of Neonatal Duodenal Atresia
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 7712
Record Dates: First submitted 2022-11-09; First posted 2023-11-02 (Actual); Last update posted 2023-12-08 (Actual); Status verified 2023-12

CONDITIONS: Congenital Duodenal Atresia
Keywords: Congenital duodenal atresia; Neonatal obstruction; Laparascopic; Laparotomy; Neonatal duodenal atresia
MeSH Terms: conditions — Familial duodenal atresia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Congenital duodenal atresia is a common cause of neonatal obstruction affecting 1 in 5000-10000 neonates. Laparoscopic management of this malformation is becoming increasingly common. However, few comparative studies exist and are often monocentric including few patients. This study will be multicentric, international and comparative to determine the place of laparoscopic surgery in the management of congenital duodenal atresia.

ELIGIBILITY:
Inclusion criteria:

* Minor subject
* Subject having undergone neonatal surgery for congenital duodenal atresia or stenosis in the different participating centers between January 2009 and December 2019
* Subject (and/or his/her parental authority) who has not expressed, after information, his/her opposition to the reuse of his/her data for the purpose of this research

Criteria for non-inclusion:

* Subject (and/or his/her parental authority) who has indicated, after information, his/her opposition to the re-use of his/her data for the purposes of this research
* Conversion linked to a renunciation of the surgeon, procedure not started (optical introduction, unfeasibility by the surgeon due to lack of experience or technical impossibility)

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Minor subject having undergone neonatal surgery for congenital duodenal atresia or stenosis in the different participating centers between January 2009 and December 2019
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2020-03-13 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
rate of complications | 3 months after laparoscopic surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Service de Chirurgie pédiatrique - CHU de Strasbourg - France, Strasbourg, France